CLINICAL TRIAL: NCT05750628
Title: A Multi-part, Multi-center PLATform Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of Anti-malarial Agents Administered as Monotherapy and/or Combination Therapy IN Patients With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Platform Study to Evaluate the Efficacy and Safety of Anti-malarial Agents in Patients With Uncomplicated Plasmodium Falciparum Malaria
Acronym: PLATINUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CADPT13A12201
Record Dates: First submitted 2023-02-17; First posted 2023-03-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: malaria; uncomplicated malaria; Plasmodium falciparum; platform study; PLATINUM
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — INE963; NITD 609; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Masking Description: This study is open-label, but certain members of the CTT will be blinded to the treatment information
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort A1: Dose Level 1 INE963 (Experimental): Cohort A1: Dose Level 1 INE963
  Interventions: Drug: INE963
- Cohort A1: Dose Level 2 INE963 (Experimental): Cohort A1: Dose Level 2 INE963
  Interventions: Drug: INE963
- Cohort A1: Dose Level 3 INE963 (Experimental): Cohort A1: Dose Level 3 INE963
  Interventions: Drug: INE963
- Cohort B1: Cipargamin + INE963 (Experimental): Cohort B1: Cipargamin + INE963
  Interventions: Drug: KAE609 (Cipargamin)
- Cohort B1: SoC (Coartem) (Active Comparator): Cohort B1: SoC (Coartem)
  Interventions: Drug: SoC (Coartem)
- Cohort B2: Cipargamin + KLU156 (Experimental): Cohort B2: Cipargamin + KLU156
  Interventions: Drug: KAE609 (Cipargamin); Drug: KLU156
- Cohort B2: SoC (Coartem) (Active Comparator): Cohort B2: SoC (Coartem)
  Interventions: Drug: SoC (Coartem)
- Cohort C2: Cipargamin + KLU156 (Experimental): Cohort C2: Cipargamin + KLU156
  Interventions: Drug: KAE609 (Cipargamin); Drug: KLU156
- Cohort C2: SoC (Coartem) (Active Comparator): Cohort C2: SoC (Coartem)
  Interventions: Drug: SoC (Coartem)
- Cohort A1: Dose Level 4 INE963 (Experimental): Cohort A1: Dose level 4 INE963
  Interventions: Drug: INE963

INTERVENTIONS:
Drug: INE963 — oral INE963
  Arms: Cohort A1: Dose Level 1 INE963; Cohort A1: Dose Level 2 INE963; Cohort A1: Dose Level 3 INE963; Cohort A1: Dose Level 4 INE963
Drug: KAE609 (Cipargamin) — oral KAE609 (Cipargamin)
  Arms: Cohort B1: Cipargamin + INE963; Cohort B2: Cipargamin + KLU156; Cohort C2: Cipargamin + KLU156
Drug: SoC (Coartem) — SoC (Coartem)
  Arms: Cohort B1: SoC (Coartem); Cohort B2: SoC (Coartem); Cohort C2: SoC (Coartem)
Drug: KLU156 — oral sachet KLU156 (KAF156 + lumefantrine)
  Arms: Cohort B2: Cipargamin + KLU156; Cohort C2: Cipargamin + KLU156

SUMMARY:
Platform study to evaluate the efficacy and safety of anti-malarial agents in patients with uncomplicated Plasmodium falciparum malaria

DETAILED DESCRIPTION:
The purpose of this platform study is to evaluate the parasiticidal effect and potential for cure with different anti-malarial agents administered as monotherapy and/or in combination therapy with other anti-malarial agents in adults, adolescents, and children with uncomplicated Plasmodium falciparum malaria. Additionally, the safety, tolerability, and pharmacokinetics of these anti-malarial agents will be evaluated for dose selection for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age for Part A, ≥12 years of age for Part B and 2 to <12 years of age for Part C at screening.
2. Patients must have acute uncomplicated P. falciparum malaria mono infection at screening confirmed by a parasite count between 5,000 to 150,000 asexual parasite count/μl of blood for P. falciparum for Part A and between 1,000 to 150,000 asexual parasite count/μl of blood for Parts B and C.
3. Patients in Part A must weigh between 40 kg and 90 kg. Patients in Part B must weigh between 35 kg and 90 kg at screening. Patients in Part C must weigh at least 10 kg at screening.
4. Axillary temperature ≥ 37.5ºC or oral/tympanic/rectal temperature ≥ 38.0ºC; or history of fever during the previous 24 hours.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria at screening or mixed Plasmodium infection (i.e., infection with more than one malaria species) at screening
2. Moderate to severe anemia, chronic hemoglobinopathy (Hemoglobin level < 8 g/dL), or known chronic underlying disease such as sickle cell disease at screening
3. Known clinically significant liver disease (e.g., chronic hepatitis, liver cirrhosis (compensated or decompensated), history of hepatitis B or C, hepatitis A or B vaccination in the last 3 months, known gallbladder or bile duct disease, acute or chronic pancreatitis. Clinical or laboratory evidence of any of the following at screening:

   * AST/ALT > 3 x the upper limit of normal range (ULN), regardless of the level of total bilirubin
   * AST/ALT > 1.5 and ≤ 2 x ULN and total bilirubin is > ULN
   * Total bilirubin > 2 x ULN, regardless of the level of AST/ALT
4. Any known/suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection at screening.
5. Pregnant or nursing (lactating) women, women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using methods of effective contraception, and sexually active patients not willing to practice effective contraception.
6. History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study such as:

   * Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
   * History of familial long QT syndrome or known family history of Torsades de Pointe.
   * Resting heart rate (physical exam or 12 lead ECG) < 50 bpm

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Part A: parasite clearance time (PCT) | up to Day 7
  Part A: To assess the parasite clearance time (PCT) of oral doses of an anti-malarial agent administered as monotherapy in patients with uncomplicated P. falciparum malaria. PCT is defined as the time from the first positive blood slide at inclusion to the time of the first negative slide followed by two consecutive slides.
Part B and C: polymerase chain reaction (PCR) corrected adequate clinical and parasitological response (ACPR) | Day 29
  Part B and C: To assess the 28-day cure rate of an anti malarial agent administered orally as combination therapy versus the standard of care (SoC) in patients with uncomplicated P. falciparum malaria. ACPR is defined as the absence of parasitemia on Study Day 29 irrespective of axillary temperature, without previously meeting any of the criteria of Early Treatment Failure (ETF) or Late Clinical Failure (LCF) or Late Parasitological Failure (LPF).

SECONDARY OUTCOMES:
Part A: PCR-corrected and uncorrected ACPR | Day 29
  Part A: To assess the 28-day cure rate of an anti malarial agent administered orally as monotherapy in patients with uncomplicated P. falciparum malaria
Parts B and C: PCT | up to Day 7
  Part B and C: To assess the parasite clearance time (PCT) of oral combinations of anti malarial agents versus the standard of care (SoC) in patients with uncomplicated P. falciparum malaria
Parts B and C: PCR-uncorrected ACPR | Day 29
  Part B and C: To assess the 28-day cure rate of an anti malarial agent administered orally as combination therapy versus the SoC in patients with uncomplicated P. falciparum malaria
Area under the concentration-time curve from time zero to the last measurable concentration sampling time (AUClast) of the anti-malarial agents (wherever possible) | Day 22
  To characterize the pharmacokinetics (PK) of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sample time (tlast)
Area under the concentration-time curve from time zero to infinity (AUCinf) of the anti-malarial agents (wherever possible) | Day 22
  To characterize PK of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. AUCinf is the AUC from time zero to infinity.
Maximum observed concentration (Cmax) of the anti-malarial agents | Day 22
  To characterize PK of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. Cmax is the maximum (peak) observed plasma, blood, serum, or other blood fluid drug concentration after single dose administration.
Time to reach maximum observed concentration (Tmax) | Day 22
  To characterize PK of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. Tmax is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration.
Elimination half-life (T1/2) of the anti-malarial agents (wherever possible) | Day 22
  To characterize PK of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. T1/2 is the elimination half-life associated with the terminal slope of a semi-logarithmic concentration-time curve.
Total body clearance (CL/F) of the anti-malarial agents (wherever possible) | Day 22
  To characterize PK of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. Cl/F is the total body clearance of drug from the plasma.
Apparent volume of distribution (V/F) of the anti-malarial agents (wherever possible) | Day 22
  To characterize PK of each anti-malarial agent administered orally as monotherapy [Part A] and/or as combination therapy [Parts B and C] in patients with uncomplicated P. falciparum malaria. V/F is the apparent volume of distribution during terminal phase.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 43
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs), and laboratory results qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Locations (12):
- Burkina Faso (2):
  - Novartis Investigative Site, Banfora
  - Novartis Investigative Site, Nanoro
- Côte d’Ivoire (2):
  - Novartis Investigative Site, Abidjan
  - Novartis Investigative Site, Azaguié
- Gabon (2):
  - Novartis Investigative Site, Lambaréné
  - Novartis Investigative Site, Libreville
- Ghana (2):
  - Novartis Investigative Site, Kintampo
  - Novartis Investigative Site, Navrango
- Kenya (2):
  - Novartis Investigative Site, Ahero, Kisumu County
  - Novartis Investigative Site, Kisumu
- Uganda (2):
  - Novartis Investigative Site, Kampala
  - Novartis Investigative Site, Tororo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.